CLINICAL TRIAL: NCT07037368
Title: Impact of Delivery Mode on Coccydynia, Pelvic Girdle Pain and Rectus Diastasis in Postpartum Females: a Comparative Study
Brief Title: Impact of Delivery Mode on Coccydynia, Pelvic Girdle Pain and Rectus Diastasis in Postpartum Females
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: DPT/Batch-Fall20/1015
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Pelvic Girdle Pain; Rectus Diastasis
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Impact of Delivery Mode
  Interventions: Behavioral: Impact of Delivery Mode

INTERVENTIONS:
Behavioral: Impact of Delivery Mode — investigates the impact of delivery mode vaginal delivery versus cesarean section on the prevalence and severity of three postpartum musculoskeletal complications: coccydynia, pelvic girdle pain (PGP), and rectus diastasis (RD). Conducted on postpartum females

SUMMARY:
This comparative observational study investigates the impact of delivery mode vaginal delivery versus cesarean section on the prevalence and severity of three postpartum musculoskeletal complications: coccydynia, pelvic girdle pain (PGP), and rectus diastasis (RD). Conducted on postpartum females aged 20-40 years within 6 weeks to 6 months after childbirth, the study aims to highlight musculoskeletal outcomes often overlooked in standard postpartum care.

DETAILED DESCRIPTION:
A total of 73 participants were selected through non-probability sampling from rehabilitation centers and home-based postpartum populations in Lahore. Pain intensity and musculoskeletal impairments were assessed using validated tools: the Visual Analog Scale (VAS) for coccydynia, Pelvic Girdle Questionnaire (PGQ) for PGP, and finger-width palpation technique for RD. The data collection involved both self-reported questionnaires and clinical assessments by trained professionals. The goal is to identify how delivery mode influences musculoskeletal health and to support the development of more tailored physiotherapy interventions and postpartum care strategies.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum females aged 20-40 years
* Females who delivered via vaginal delivery or cesarean section
* 6 weeks to 6 months postpartum period
* Willingness to participate and provide informed consent

Exclusion Criteria:

* Females with a history of pelvic or spinal surgery prior to pregnancy
* Known cases of pre-existing musculoskeletal disorders (e.g., scoliosis, chronic back pain)
* Multiple pregnancies (twins or more) in the current or previous delivery
* Postpartum complications unrelated to delivery mode (e.g., sepsis, trauma)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This comparative observational study investigates the impact of delivery mode vaginal delivery versus cesarean section on the prevalence and severity of three postpartum musculoskeletal complications: coccydynia, pelvic girdle pain (PGP), and rectus diastasis (RD).
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | 6 Month
  A 10 cm horizontal line marked from 0 (no pain) to 10 (worst imaginable pain). Scoring: The participant marks a point on the line that best represents their pain intensity. The score is measured in centimeters from the "no pain" end. Higher scores indicate more severe pain.
Pelvic Girdle Questionnaire (PGQ) | 6 Months
  Contains 25 items divided into two domains: activity limitations (20 items) and symptoms (5 items).
  Scoring: Each item is rated on a 4-point scale (0 = not at all, 1 = to a small extent, 2 = to some extent, 3 = to a great extent). Scores are summed, converted into a percentage of the maximum possible score. Higher percentages reflect greater pelvic girdle pain and disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Superior University CRC, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No